CLINICAL TRIAL: NCT01719562
Title: Improving Exercise Capacity With a Tailored Physical Activity Intervention in Lymphoma and Breast Cancer Patients Undergoing Treatment - An Addendum to NIH R01CA167821 "Early Imaging Detection of Cardiovascular Injury After Cancer"
Brief Title: MRI in Detecting Heart Damage in Patients With Cancer Receiving Chemotherapy With Exercise Capacity Addendum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00020968; NCI-2012-01613 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA012197 (NIH); CCCWFU 99112 (Other: Wake Forest University Health Sciences); R01CA167821 (NIH); R21CA226960 (NIH)
Record Dates: First submitted 2012-10-11; First posted 2012-11-01 (Estimated); Results first posted 2023-05-16 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Cardiac Toxicity; Malignant Neoplasm; Breast Cancer
MeSH Terms: conditions — Cardiotoxicity; Neoplasms; Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy; Exercise; Exercise Test

STUDY DESIGN:
Intervention Model Description: For the exercise capacity portion of this trial, participants will be randomized to 1 of 2 arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- ADDENDUM: Physical Activity Intervention (Experimental): Participants will be offered one to two training sessions per week at onsite rehab facilities and 1-2 sessions per week at home consisting of slow 15 minute aerobic warm-up followed by 20 minutes of strength training, 15 minutes of progressive intensity aerobic exercise and 10 minute cool down.
  Interventions: Procedure: Magnetic resonance imaging; Other: Physical Activity; Device: Cardiopulmonary Exercise Testing (CPET); Other: Questionnaire Administration
- ADDENDUM: Healthy Living Instruction Group (Control Arm) (Experimental): Organized various health workshops lasting for 60 minutes to match the number of visits to the rehab centers for participants in Arm 1 with 2 sessions offered per month onsite and remaining sessions offered over the phone for 6 months. .
  Interventions: Procedure: Magnetic resonance imaging; Other: Healthy Living; Device: Cardiopulmonary Exercise Testing (CPET); Other: Questionnaire Administration
- MRI (Diagnostic) (Experimental): Patients undergo MRI scans for LV function, T1 myocardial signal, and aortic PWV at baseline, 3 months, and 24 months.
  Interventions: Procedure: Magnetic resonance imaging; Other: Physical Activity; Other: Healthy Living

INTERVENTIONS:
Procedure: Magnetic resonance imaging — Patients undergo MRI scans for left ventricular function, T1 myocardial signal, and aortic PWV at baseline, 3 months, and 24 months.
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging
Other: Physical Activity — Tailored aerobic exercise program onsite and at home.
  Arms: ADDENDUM: Physical Activity Intervention; MRI (Diagnostic)
Other: Healthy Living — Healthy living presentations at a centralized meeting place and over the phone.
  Arms: ADDENDUM: Healthy Living Instruction Group (Control Arm); MRI (Diagnostic)
Device: Cardiopulmonary Exercise Testing (CPET) — Performed on the treadmill using the Bruce or Modified Bruce protocol based on current fitness level.
  Arms: ADDENDUM: Healthy Living Instruction Group (Control Arm); ADDENDUM: Physical Activity Intervention
Other: Questionnaire Administration — A self-administered 13-item scale to assess fatigue in participants
  Arms: ADDENDUM: Healthy Living Instruction Group (Control Arm); ADDENDUM: Physical Activity Intervention

SUMMARY:
This trial studies how well magnetic resonance imaging (MRI) works in detecting heart damage in patients with cancer receiving chemotherapy. Diagnostic procedures, such as MRI, may help doctors predict whether patients will have heart damage caused by chemotherapy in patients with cancer receiving chemotherapy.

Exercise Capacity Addendum Brief Summary: This study is designed to demonstrate feasibility of performing the physical activity intervention and the primary outcome measures before, during and six months after initiating Anth-bC for treatment of non- or Hodgkin lymphoma. This study will test the potential for a novel (lifestyle) intervention designed to improve exercise capacity, health-related quality of life and cardiac and cognitive dysfunction. This data will inform the development of the R33 phase of the clinical trial to determine if the physical activity intervention can reduce exercise intolerance in this high-risk population. In addition, cardiac MRI data from individuals within this pilot will be compared to cardiac MRI data from individuals in the parent study that did not undergo either of the two interventional arms of this study.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To design an automated MRI hardware/software platform for measuring and reporting left ventricular (LV) function (volumes, strain, and ejection fraction [EF]), T1 myocardial signal, and aortic pulse wave velocity (PWV).

II. To determine if pre- to 3 month post-anthracycline-based chemotherapy (Anth-bC) changes in our MRI platform generated measures of LV volumes, EF, strain, myocardial T1, and aortic PWV predict pre- to 24 month post-Anth-bC differences in these same parameters.

OUTLINE:

Patients undergo MRI scans for LV function, T1 myocardial signal, and aortic PWV at baseline, 3 months, and 24 months.

Exercise Capacity Addendum Objectives:

Primary Objective:

* To provide critical participant enrollment data necessary to accomplish the R01 submission, including:
* Feasibility of screening, enrolling, and randomizing 21 Non or Hodgkin lymphoma and stage I-IV breast cancer patients including the reasons for failed randomization,
* Identification of barriers for participating in, or adhering to the Patient ES-AI and the Healthy Living Control Group.

Secondary Objective:

• In these 21 patients, at study initiation then 3 and 6 months after initiating Anth-bC or other potentially cardiotoxic cancer therapies, to assess the ability to ascertain: peak exercise cardiac output, calculated arteriovenous oxygen difference (A-V O2) and VO2 (maximum rate of oxygen), and pre-exercise measures of left ventricular and cognitive function, health-related quality of life, six-minute walk distance (6min WD) and fatigue. Ascertainment of the left ventricular function and health-related rate quality of life will be attempted in a manner similar to ascertainment of these variables from 47 individuals with lymphoma in the parent study.

ELIGIBILITY:
PARENT STUDY:

Inclusion Criteria:

* Receiving >= 350 mg/m^2 of Anth-bC therapy, or a combination of Anth-bC (>= 250 mg/m^2) and subsequent paclitaxel or Herceptin
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Intracranial metal, pacemakers, defibrillators, functioning neurostimulator devices, or other implanted electronic devices
* Ferromagnetic cerebral aneurysm clips, or other intraorbital/intracranial metal
* Allergy to gadolinium or other severe drug allergies
* Unstable angina
* Significant ventricular arrhythmias (> 20 premature ventricular contractions [PVCs]/minute due to gating difficulty)
* Acute myocardial infarction within 28 days
* Atrial fibrillation with uncontrolled ventricular response
* Moderate or severe aortic stenosis
* Claustrophobia
* Congestive heart failure (New York Heart Association [NYHA] class III or IV)
* Significant valvular disease, or significant pulmonary disease requiring supplemental oxygen therapy
* Participants unwilling to complete the protocol (24 month duration)
* Women who are pregnant
* Patients unable or unwilling to provide informed consent

EXERCISE CAPACITY ADDENDUM:

Inclusion Criteria:

* Men and women aged 18-85 with non- or Hodgkin lymphoma or I-IV stage breast cancer patients that expect to receive an anthracycline based chemotherapeutic regimen or other potentially cardiotoxic cancer therapies (e.g. chemotherapy regimens [anthracyclines, trastuzumab]), immuno-therapies (immune checkpoint inhibitors [ICI's]) or radiation (within 8 weeks of completion).
* Potential enrollees will need the capacity to walk at least two (2) city blocks on a flat surface.
* English speaking participants only will be enrolled.
* Stage IV breast cancer participants must have a 2 year survival prognosis and approval from their physician.

Exclusion Criteria: The following are relative contraindications and can be considered by the medical director of the study:

* Uncontrolled hypertension (systolic blood pressure >190 mm Hg or diastolic blood pressure >100 mm Hg)
* A recent history of alcohol or drug abuse.
* Inflammatory conditions such as lupus or inflammatory bowel disease, or another medical condition that might compromise safety or successful completion.
* Other exclusions include those with contraindications to MRI such as ferromagnetic cerebral aneurysm clips or other intracranial metal, pacemakers, defibrillators, functioning neurostimulator devices or other implanted electronic devices.
* Unstable angina.
* Inability to exercise on a treadmill or stationary cycle.
* Significant ventricular arrhythmias (>20 PVCs/min due to gating difficulty).
* Atrial fibrillation with uncontrolled ventricular response.
* Acute myocardial infarction within 28 days.
* Moving within 12 months of enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Hundley, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina
  - Virginia Commonwealth University Health Sciences, Richmond, Virginia

REFERENCES:
- [Derived] Costa JV, Lucas AR, Mihalko SL, Brubaker PH, Marshall A, Leitzelar B, Wolle BR, Norton S, Franco RL, Via J, Yazbeck V, Vaidya R, Seegars MB, D'Agostino R Jr, Wagner L, Hundley WG. Feasibility and preliminary efficacy of a physical activity intervention in adults with lymphoma undergoing treatment. Pilot Feasibility Stud. 2025 Jan 14;11(1):6. doi: 10.1186/s40814-024-01580-7. PMID 39810280
- [Derived] Mabudian L, Reding K, D'Agostino RB Jr, Heiston EM, Bellissimo MP, Olson K, Ntim WO, Klepin HD, Dressler EV, Moore T, Jordan JH, O'Connell NS, Ladd A, Weaver KE, Ky B, Wagner LI, Hackney MH, Lesser GJ, Hundley WG; UPBEAT Study Team. The relationship between body composition and left ventricular performance in women with breast, lymphoma, or sarcoma cancer. Cardiooncology. 2024 Jun 6;10(1):34. doi: 10.1186/s40959-024-00233-1. PMID 38845066
- [Derived] Garg R, D'Agostino RB Jr, O'Connell N, Lesser GJ, Salloum FN, Hines AL, Melendez GC, Jordan JH, Ky B, Wagner LI, Sutton AL, Bottinor W, Olson KC, Ladd AC, Hundley WG; UPBEAT Study Team. Hypertension Severity and Declines in Left Ventricular Ejection Fraction Among Women Receiving Adjuvant Chemotherapy for Breast Cancer (WF-97415 UPBEAT). Hypertension. 2024 Jun;81(6):1365-1373. doi: 10.1161/HYPERTENSIONAHA.123.21817. Epub 2024 Apr 18. PMID 38634292

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ADDENDUM: Physical Activity Intervention | ADDENDUM: Healthy Living Instruction Group (Control Arm)
Started | 20 | 8
Completed | 17 | 8
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 1 | 0
Not completed — New cancer diagnosis | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ADDENDUM: Physical Activity Intervention | ADDENDUM: Healthy Living Instruction Group (Control Arm) | Total
Number analyzed (Participants) | 20 | 8 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (16.8) | 56.8 (12.7) | 53.65 (16.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 4 | 18
  Male | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 17 | 6 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 8 | 28
Diagnosis: Hodgkin Lympoma, Non-Hodgkin Lymphoma, Breast Cancer [Count of Participants; unit: Participants]
  Hodgkin Lymphoma | 7 | 4 | 11
  Non-Hodgkin Lymphoma | 6 | 3 | 9
  Breast Cancer | 7 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completing the Trial (Exercise Capacity Addendum)
Description: The number of participants who completed the intervention.
Time Frame: 6 months after treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | ADDENDUM: Physical Activity Intervention | ADDENDUM: Healthy Living Instruction Group (Control Arm)
Number analyzed (Participants) | 20 | 8
Participants | 17 | 8

2. Primary Outcome: Number of Participants Able to Complete Assessments (Exercise Capacity Addendum)
Description: Number of participants who completed the 6-minute walk test at 6-months.
Time Frame: 6 months after treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | ADDENDUM: Physical Activity Intervention | ADDENDUM: Healthy Living Instruction Group (Control Arm)
Number analyzed (Participants) | 20 | 8
Participants | 14 | 7

3. Secondary Outcome: Peak Exercise Cardiac Output (Exercise Capacity Addendum)
Description: Peak exercise cardiac output refers to the amount of blood that the heart pumps out per minute. It is an important measure of how effectively the heart is working to deliver oxygen and nutrients to the body's tissues. Peak exercise cardiac output was measured in a cardiac magnetic resonance imaging (MRI) exam.
Time Frame: 6 months after treatment
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | ADDENDUM: Physical Activity Intervention | ADDENDUM: Healthy Living Instruction Group (Control Arm)
Number analyzed (Participants) | 8 | 6
mL/min | 16900 (3350) | 15700 (4100)

4. Secondary Outcome: Arteriovenous Oxygen Difference (A-V O2) (Exercise Capacity Addendum)
Description: Arteriovenous Oxygen Difference (A-V O2) is the difference in oxygen levels between arterial blood and venous blood. A-V O2 difference is important because it reflects how much oxygen is being used by the body's tissues during exercise or physical activity. A higher A-V O2 difference is generally considered better.
Time Frame: 6 months after treatment initiation
Population: Hospital restrictions due to COVID-19 prevented the data collection of A-V O2 on all participants who completed the study.
Measure: Mean (Standard Deviation); unit: mL/100 mL
Arm/Group | ADDENDUM: Physical Activity Intervention | ADDENDUM: Healthy Living Instruction Group (Control Arm)
Number analyzed (Participants) | 8 | 6
mL/100 mL | 0.00182 (0.000322) | 0.00150 (0.000362)

5. Secondary Outcome: Maximum Rate of Oxygen Consumption (VO2) (Exercise Capacity Addendum)
Description: Maximum rate of oxygen consumption (VO2) is an objective measure of cardiorespiratory fitness. VO2 was assessed with a cardiopulmonary exercise test (CPET). Higher VO2 represents greater cardiorespiratory fitness.
Time Frame: 6 months after treatment initiation
Population: Hospital restrictions due to COVID-19 prevented the data collection of VO2 on all participants who completed the study.
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | ADDENDUM: Physical Activity Intervention | ADDENDUM: Healthy Living Instruction Group (Control Arm)
Number analyzed (Participants) | 9 | 6
mL/kg/min | 29.6 (5.83) | 23.6 (10.2)

6. Secondary Outcome: Left Ventricular Function (Exercise Capacity Addendum)
Description: Left ventricular ejection fraction (LVEF, %) is a measure of cardiac function. LVEF was assessed with a cardiac magnetic resonance imaging (MRI) exam. The higher the LVEF, the more efficiently the heart is at pumping blood to the rest of the body with every heart beat.
Time Frame: 6 months after treatment initiation
Population: Hospital restrictions due to COVID-19 prevented the data collection of LVEF on all participants who completed the study.
Measure: Mean (Standard Deviation); unit: LVEF Percentage
Arm/Group | ADDENDUM: Physical Activity Intervention | ADDENDUM: Healthy Living Instruction Group (Control Arm)
Number analyzed (Participants) | 9 | 6
LVEF Percentage | 65.3 (8.06) | 65.1 (5.76)

7. Secondary Outcome: Cognitive Function- Controlled Oral Word Association (COWA) Test (Exercise Capacity Addendum)
Description: The COWA test was used to assess cognitive function and verbal fluency. Participants were asked to produce as many words as they can that begin with the given letter (i.e. T or L) within a 1-min time period. The COWA test total score was measured by summing the total number of acceptable words produced for three different letters. Minimum possible score for the COWA text is 0. There is no maximum possible score. Higher scores represent greater verbal fluency.
Time Frame: 6 months after treatment initiation
Population: Hospital restrictions due to COVID-19 prevented the data collection of the COWA test on all participants who completed the study.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ADDENDUM: Physical Activity Intervention | ADDENDUM: Healthy Living Instruction Group (Control Arm)
Number analyzed (Participants) | 14 | 4
Scores on a scale | 46.5 (9.53) | 39.3 (10.6)

8. Secondary Outcome: Health-Related Quality of Life (Exercise Capacity Addendum)
Description: The Functional Assessment of Cancer Treatment-Lymphoma (FACT-Lym) is a 42-item scale used to assess the health-related quality of life of lymphoma survivors. The FACT-Lym questionnaire examines the four primary domains of HRQL: physical, social, emotional, and functional well-being, and patient's concerns related to lymphoma. The FACT-Lym was examined as a total score, ranging from 0 to 168 points. Higher scores reflect better health-related quality of life.
Time Frame: 6 months after treatment initiation
Population: Some participants refused or failed to complete the FACT-Lym survey at 6-months.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ADDENDUM: Physical Activity Intervention | ADDENDUM: Healthy Living Instruction Group (Control Arm)
Number analyzed (Participants) | 12 | 5
Scores on a scale | 87.3 (10.3) | 76.6 (13.4)

9. Secondary Outcome: 6-minute Walk Distance (Exercise Capacity Addendum)
Description: The 6-minute walk test is a low cost sub-maximal exercise test that serves as an indirect measure of cardiorespiratory fitness. Participants were instructed to walk at their own pace to cover as much ground (in meters) as possible for 6 minutes.
Time Frame: 6 months after treatment initiation
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | ADDENDUM: Physical Activity Intervention | ADDENDUM: Healthy Living Instruction Group (Control Arm)
Number analyzed (Participants) | 14 | 7
meters | 543 (90.6) | 457 (77.0)

10. Secondary Outcome: Functional Assessment of Cancer Therapy - (FACT-Fatigue) (Exercise Capacity Addendum)
Description: The FACT-fatigue is a 13-item scale that has been widely used to assess cancer-related fatigue. The FACT-fatigue questionnaire was scored by summing all 13 items with a reverse point system. This produces a range of 0 to 52, with a higher score indicating better functioning and less fatigue.
Time Frame: 6 months after treatment initiation
Population: Some participants refused or failed to complete the FACT-Fatigue survey at 6-months.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ADDENDUM: Physical Activity Intervention | ADDENDUM: Healthy Living Instruction Group (Control Arm)
Number analyzed (Participants) | 15 | 8
Scores on a scale | 42.0 (6.20) | 32.4 (8.52)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | ADDENDUM: Physical Activity Intervention | ADDENDUM: Healthy Living Instruction Group (Control Arm)
All-Cause Mortality (participants affected / at risk) | 1/20 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/8
Other Adverse Events (participants affected / at risk) | 1/20 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADDENDUM: Physical Activity Intervention (N=20) | ADDENDUM: Healthy Living Instruction Group (Control Arm) (N=8)
Nausea due to home-based exercise session (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant experienced nausea during online kickboxing class. Recovered within 2 hours after exercise. Adjusted exercise recommendation to stay below high HR ranges. Participant completed the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT01719562/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/62/NCT01719562/ICF_000.pdf